CLINICAL TRIAL: NCT05077852
Title: Intravesical Prostatic Protrusion Mimicking Urothelial Cell Carcinoma of the Bladder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: IPP-BC
Record Dates: First submitted 2021-10-12; First posted 2021-10-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Bladder Cancer; Benign Prostatic Hyperplasia; Hematuria
Keywords: Bladder cancer; Benign prostatic hyperplasia; Hematuria; Ultrasonography
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Hyperplasia; Hematuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystoscopy Bladder Cancer: Patients diagnosed with primary bladder cancer at the base, trigone or neck of the bladder by cystoscopy.
  Interventions: Diagnostic Test: Urethrocystoscopy
- Cystoscopy IPP: Patients diagnosed with intravesical prostate protrusion (IPP) at the base, trigone or neck of the bladder by cystoscopy.
  Interventions: Diagnostic Test: Urethrocystoscopy

INTERVENTIONS:
Diagnostic Test: Urethrocystoscopy — Patients diagnosed with a primary bladder cancer at the base, trigone or neck of the bladder with USG in the urology clinic will be evaluated with urethrocystoscopy. With urethrocystoscopy, patients definitive diagnosed with bladder cancer and IPP.

SUMMARY:
In this study, investigators aim to determine the true positivity of bladder cancer identified in the bladder base, trigone or neck on ultrasonography (USG) in patients presenting with hematuria or lower urinary tract symptoms, by confirming with the gold standard cystoscopy and biopsy results. It also aims to explore criteria that would allow to differentiate between intravesical prostate protrusion (IPP) due to benign prostatic hyperplasia (BPH) and bladder cancer indicated at the bladder floor, trigone and neck by evaluating false positive results.

DETAILED DESCRIPTION:
The most common symptom in bladder cancer is hematuria, although the rate of bladder cancer is 18.9% in patients presenting with gross hematuria and 4.8% in patients presenting with microscopic hematuria. For this reason, unnecessary and invasive procedures are applied to most of the patients investigated. USG is considered the first-line imaging technique in the evaluation of upper and lower urinary tract disease. It is a non-invasive technique that does not involve ionizing radiation, and can be used in the evaluation of kidney, prostate and bladder anatomy. In addition, USG is used to evaluate malignant tumors of the urinary system or benign causes such as BPH, urinary tract stones that may cause hematuria. Cystoscopy is the gold standard test for diagnosing bladder cancer, but cystoscopy causes discomfort and can carry risks such as infection and bleeding. Suspicious findings as a result of USG imaging may lead to more invasive tests such as cystoscopy. An example of this is performing a biopsy under general anesthesia to confirm a positive or negative finding. The annual costs of these examinations, which emerge as further examinations as a result of incorrect evaluations, are important. In England, patients with hematuria and normal investigation cost the National Health Service £33.5 million in one year.

IPP, or median lobe, is a phenomenon in which the prostate adenoma expands into the bladder along the plane of lowest resistance. IPP originating from the base of the prostate may enlarge and protrude into the bladder and form a regional lesion on the neck, trigone and posterior wall of the bladder. IPP cannot be detected adequately by conventional digital rectal examination (DRE), nor can it be diagnosed with sufficient accuracy by examinations such as noninvasive USG. In the literature, some studies evaluated the diagnosis of IPP by USG, and the full spectrum of IPP was not defined due to the scarcity of clinical series. IPP is seen as protruding structures within the bladder in the coronal plane of USG and can be easily misdiagnosed as a bladder-derived lesion. Thus, IPP, which is a manifestation of BPH, located at the base of the prostate and extending into the bladder, can easily be misdiagnosed as bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Hematuria
* Patients diagnosed with primary bladder cancer at the base, trigone or neck of the bladder by USG.

Exclusion Criteria:

* Previous history of urinary tract tumor
* Chronic kidney disease
* Use of antimuscarinic drugs
* Active urinary tract infection
* Bladder stone
* Previous history of lower urinary tract surgery or urethral stricture

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with primary bladder cancer at the base, trigone or neck of the bladder by USG.
Sampling Method: Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of a positive screening test truly have the bladder cancer | 3 months
  Rate of a positive screening test truly have the bladder cancer in patients who diagnosed with bladder cancer at the base, trigone or neck by USG

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khadhouri S, Gallagher KM, MacKenzie K, Shah TT, Gao C, Moore S, Zimmermann E, Edison E, Jefferies M, Nambiar A, MacLennan G, McGrath JS, Kasivisvanathan V; IDENTIFY Protocol Collaborators Group. IDENTIFY: The investigation and detection of urological neoplasia in patients referred with suspected urinary tract cancer: A multicentre cohort study. Int J Surg Protoc. 2020 Feb 28;21:8-12. doi: 10.1016/j.isjp.2020.02.002. eCollection 2020. PMID 32322764
- [Background] Gandhi J, Weissbart SJ, Kim AN, Joshi G, Kaplan SA, Khan SA. Clinical Considerations for Intravesical Prostatic Protrusion in the Evaluation and Management of Bladder Outlet Obstruction Secondary to Benign Prostatic Hyperplasia. Curr Urol. 2018 Oct;12(1):6-12. doi: 10.1159/000447224. Epub 2018 Jun 30. PMID 30374274
- [Background] Chang SS, Boorjian SA, Chou R, Clark PE, Daneshmand S, Konety BR, Pruthi R, Quale DZ, Ritch CR, Seigne JD, Skinner EC, Smith ND, McKiernan JM. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline. J Urol. 2016 Oct;196(4):1021-9. doi: 10.1016/j.juro.2016.06.049. Epub 2016 Jun 16. PMID 27317986